CLINICAL TRIAL: NCT07322055
Title: A Correlational Study Between Genetic Profiles and Clinical Characteristics in Subjects With Disruptive Behavior Disorder Diagnosis, With or Without Callous-Unemotional Traits.
Brief Title: Genetic and Clinical Correlates of Disruptive Behavior Disorder With and Without Callous-Unemotional Traits
Acronym: GENCU 2025
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS Fondazione Stella Maris (Other)
Collaborators: University of Pisa (Other)
Responsible Party: Sponsor
Other Study IDs: GENCU 2025
Record Dates: First submitted 2025-12-22; First posted 2026-01-07 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-12

CONDITIONS: Conduct Disorder; Oppositional Defiant Disorder; Callous Unemotional Traits
Keywords: Conduct Disorder; Oppositional Defiant Disorder; Callous Unemotional Traits; Genetics
MeSH Terms: conditions — Conduct Disorder; Oppositional Defiant Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Each participant has provided a non-invasive saliva sample using a self-collection kit. The samples have been processed to extract genomic DNA, which is stored securely at -20°C.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Disruptive Behavior Disorders (DBD), such as Conduct Disorder (CD) and Oppositional Defiant Disorder (ODD), affect children and adolescents in different ways. Research has shown that some individuals with DBD also display callous-unemotional (CU) traits, including a lack of guilt, uncaring behavior, and shallow emotions. This subgroup tends to have more severe symptoms and a higher risk of negative outcomes.

Previous studies suggest that genetic factors may play a role in the development of DBD with CU traits. For example, specific variations of the MAOA gene have been linked to difficulties in recognizing and processing emotions such as sadness and fear, which are often impaired in individuals with CU traits.

This study aims to explore how broader genetic profiles may affect DBD and CU traits. In the already enrolled sample, we will explore correlations between the collected clinical data and a larger set of genetic variants. The goal is to improve knowledge about the genetic factors that contribute to differences in behavior, which may help inform strategies to identify risk and resilience in individuals with disruptive behavioral traits.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of Conduct Disorder or Oppositional Defiant Disorder, obtained using the Kiddie Schedule for Affective Disorders and Schizophrenia-Present and Lifetime version (K-SADS-PL);
* Age 7-16 years;
* Intelligence Quotient > 85;
* Italian nationality and Caucasian ethnicity (excluding Sardinians for reasons of ethnic uniformity);
* No relatives already enrolled in the study.

Exclusion Criteria:

* Lack of signed Informed Consent;
* Diagnosis of Pervasive Developmental Disorder according to K-SADS-PL.

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population consists of children and adolescents aged 7-16 years diagnosed with Conduct Disorder or Oppositional Defiant Disorder and treated at a specialized outpatient clinic for childhood behavioral disorders.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-10-07 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Callous-unemotional traits - ICU | At baseline
  Callous-unemotional (CU) traits are assessed using the child-report Inventory of Callous-Unemotional Traits (ICU), a 24-item questionnaire measuring Callousness, Uncaring, and Unemotional traits. Answers are rated on a 4-point Likert scale (0 = Not at All True, 3 = Definitely True). Total score range is 0 to 72, with higher scores indicating more prominent CU traits.
Callous-unemotional traits - APSD | At baseline
  Callous-unemotional traits are assessed with the Callous-Unemotional (CU) subscale of the child-report Antisocial Process Screening Device (APSD). The CU subscale includes 6 items rated on a 3-point Likert scale (0 = Not at All True, 1 = Sometimes True, 2 = Definitely True). Scores range from 0 to 12, with higher scores suggesting higher CU traits.
Psychopathic traits | At baseline
  Psychopathic traits are assessed with the Self-Report Psychopathy Scale, Fourth Edition (SRP-4), which provides scores across four dimensions (Interpersonal, Affective, Lifestyle, Antisocial) and a Total score, with item responses on a 5-point Likert scale, with higher scores indicating more psychopathic traits.
Emotion processing | At baseline
  Emotion processing is evaluated by recording gaze pattern using a binocular eye-tracking system, while children are presented with emotional stimuli on a computer screen.

SECONDARY OUTCOMES:
Externalizing Problems | At baseline
  Externalizing problems are assessed using the self-report version of the Strengths and Difficulties Questionnaire (SDQ), a 25-item questionnaire. The composite Externalizing problems score is the sum of the Hyperactivity-Inattention and Conduct Problems scales. Items are rated on a 3-point Likert scale (0 = Not True, 1 = Somewhat True, 2 = Certainly True). Higher scores indicate higher externalizing problems (range 0-20).
Internalizing Problems | At baseline
  Internalizing problems are assessed using the self-report version of the Strengths and Difficulties Questionnaire (SDQ), a 25-item questionnaire. The composite Internalizing problems score is the sum of the Emotional Symptoms and Peer Problems scales. Items are rated on a 3-point Likert scale (0 = Not True, 1 = Somewhat True, 2 = Certainly True). Higher scores indicate higher internalizing problems (0-20).
Prosocial Behavior | At baseline
  Prosocial behavior are assessed using the self-report version of the Strengths and Difficulties Questionnaire (SDQ), a 25-item questionnaire. The Prosocial scale includes 5 items rated on a 3-point Likert scale (0 = Not True, 1 = Somewhat True, 2 = Certainly True). Higher scores indicate more prosocial behavior (range 0-10).
Parenting | At baseline
  Parenting practices are assessed using the parent-report Alabama Parenting Questionnaire (APQ), a 42-item questionnaire. The APQ includes five subscales: Positive Involvement, Supervision/Monitoring, Discipline Practices, Consistency, and Corporal Punishment. Higher scores indicate higher levels of the respective parenting practices.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Università di Pisa, Pisa, Pisa
  - IRCCS Fondazione Stella Maris, Pisa, Pisa